CLINICAL TRIAL: NCT05435261
Title: Ganga Hospital Scoring System In Gustilo And Anderson Classification System Type-IIIA/B Open Tibial Fractures
Brief Title: Ganga Hospital Scoring System In Type-IIIA/B Open Tibial Fractures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Abdelkarem, Director, Assiut University
Other Study IDs: GHS
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Fractures, Open
MeSH Terms: conditions — Fractures, Open | interventions — Debridement; Salvage Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: with a score below 14
  Interventions: Procedure: Debridement with Ex_Fix (salvage)
- Group II: with a score above 14
  Interventions: Procedure: BKA

INTERVENTIONS:
Procedure: BKA — Below Knee Amputation:
  * Under spinal anesthesia
  * BKA
  * closure in layers (terminal closure) with suction drain.
  Groups: Group II
Procedure: Debridement with Ex_Fix (salvage) — Debridement and External Fixation (salvage):
  * Under spinal anesthesia
  * wound debridement and wash.
  * external fixation.
  Groups: Group I

SUMMARY:
The aim of this study is to assess interobserver reliability, sensitivity for amputation, and specificity for salvage of GHS in type-III injuries with open tibial fractures and predict the potential number of inpatient days, secondary procedures that would be required, and the rate of infection

DETAILED DESCRIPTION:
Open fractures are usually high-energy injuries that can lead to life-threatening multiple injuries. It is classified as an orthopaedic emergency, and successful treatment depends on a thorough assessment and prompt treatment of the patient and wound. With the rise in severe open tibia injuries, an ideal scoring system with high specificity and sensitivity for predicting limb salvage is required. A misdiagnosis can lead to unnecessary amputations or salvage operations. A variety of scoring methods have been described for limb salvaging. The Gustilo and Anderson classification system is still the most used. Following the original classification, typeIII injuries were subdivided into type-IIIA, which denoted adequate soft-tissue coverage of the fracture despite extensive skin loss, type-IIIB, which denoted extensive soft-tissue loss, periosteal stripping, and bone exposure; and type-IIIC, which denoted an open fracture with an associated arterial injury that required repair. It has the limitations of a low intra and inter-observer agreement rate, low specificity and sensitivity to salvage and ambulation, and an inability to predict functional results in the care of Type IIIB injuries. The Ganga Hospital Score (GHS) is an open injury score developed from a high-volume trauma center that treats more than 600 open lower-limb fractures each year, far higher than a typical major trauma center in the United Kingdom. Following three clinical trials, the score was developed and has been shown to accurately predict whether a limb can be saved or must be amputated. The scoring system's nature, which takes into account particular injuries to the bone, skin, and musculotendinous units, as well as comorbid factors, has also been expanded to advise wound treatment. In medicine, scoring systems are used to rate the severity of an illness, predict the outcome, and aid in management decisions. In open injuries, an ideal score would have a sensitivity of 100%, with all limbs requiring amputation scoring at or above the threshold value, and a specificity of 100%, with all limbs that can be preserved scoring below the threshold value. Because these injuries are frequently complex clinical conditions, this is challenging to achieve. Although it is preferable to err on the side of high specificity such that only a small percentage of salvageable limbs score over the amputation threshold, high sensitivity is also necessary to limit the number of secondary amputations.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged more than 17 years
* open fractures of the tibia irrespective of the fracture site, presenting within 24 h of injury type-IIIA/B

Exclusion Criteria:

* Patients with Gustilo and Anderson types I, II, and IIIC injuries.
* complete traumatic amputations.
* patients who had initial debridement at an outside hospital.
* those with an age group less than 17 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: trauma patient with open tibial fractures type-IIIA/B
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity GHS in type- IIIA/B open tibial fractures | one year
  salvage with score below 14 and Amputation with score above 14

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mohamadean Mohamed, Professor, Study Chair — Prof. Dr; Hossam Mohamed Abubeih, Assistant Professor, Study Director — Ass. Prof. Dr

REFERENCES:
- [Background] Griffin M, Malahias M, Khan W, Hindocha S. Update on the management of open lower limb fractures. Open Orthop J. 2012;6:571-7. doi: 10.2174/1874325001206010571. Epub 2012 Nov 30. PMID 23248730
- [Background] Gustilo RB, Anderson JT. Prevention of infection in the treatment of one thousand and twenty-five open fractures of long bones: retrospective and prospective analyses. J Bone Joint Surg Am. 1976 Jun;58(4):453-8. PMID 773941
- [Background] Kumar KN, Shivanna HYS, Kumar TNS, Pratheeksh. Assessment of Ganga Hospital Open Injury Severity Score of Limbs. J Emerg Trauma Shock. 2020 Oct-Dec;13(4):317-318. doi: 10.4103/JETS.JETS_68_20. Epub 2020 Dec 7. No abstract available. PMID 33897152
- [Background] Rajasekaran S, Naresh Babu J, Dheenadhayalan J, Shetty AP, Sundararajan SR, Kumar M, Rajasabapathy S. A score for predicting salvage and outcome in Gustilo type-IIIA and type-IIIB open tibial fractures. J Bone Joint Surg Br. 2006 Oct;88(10):1351-60. doi: 10.1302/0301-620X.88B10.17631. PMID 17012427
- [Background] Rajasekaran S, Sabapathy SR. A philosophy of care of open injuries based on the Ganga hospital score. Injury. 2007 Feb;38(2):137-46. doi: 10.1016/j.injury.2006.04.135. Epub 2006 Sep 6. PMID 16950263
- [Background] Al-Hourani K, Stoddart M, Khan U, Riddick A, Kelly M. Orthoplastic reconstruction of type IIIB open tibial fractures retaining debrided devitalized cortical segments: the Bristol experience 2014 to 2018. Bone Joint J. 2019 Aug;101-B(8):1002-1008. doi: 10.1302/0301-620X.101B8.BJJ-2018-1526.R2. PMID 31362546
- [Background] Messner J, Johnson L, Taylor DM, Harwood P, Britten S, Foster P. Treatment and functional outcomes of complex tibial fractures in children and adolescents using the Ilizarov method. Bone Joint J. 2018 Mar 1;100-B(3):396-403. doi: 10.1302/0301-620X.100B3.BJJ-2017-0863.R1. PMID 29589503
- [Background] Venkatadass K, Grandhi TSP, Rajasekaran S. Use of Ganga Hospital Open Injury Severity Scoring for determination of salvage versus amputation in open type IIIB injuries of lower limbs in children-An analysis of 52 type IIIB open fractures. Injury. 2017 Nov;48(11):2509-2514. doi: 10.1016/j.injury.2017.09.010. Epub 2017 Sep 12. PMID 28918873
- [Background] Shanmuganathan R. The utility of scores in the decision to salvage or amputation in severely injured limbs. Indian J Orthop. 2008 Oct;42(4):368-76. doi: 10.4103/0019-5413.43371. PMID 19753223
- [Background] Rajasekaran S, Sabapathy SR, Dheenadhayalan J, Sundararajan SR, Venkatramani H, Devendra A, Ramesh P, Srikanth KP. Ganga hospital open injury score in management of open injuries. Eur J Trauma Emerg Surg. 2015 Feb;41(1):3-15. doi: 10.1007/s00068-014-0465-9. Epub 2014 Nov 6. PMID 26038161
- [Background] Durham RM, Mistry BM, Mazuski JE, Shapiro M, Jacobs D. Outcome and utility of scoring systems in the management of the mangled extremity. Am J Surg. 1996 Nov;172(5):569-73; discussion 573-4. doi: 10.1016/S0002-9610(96)00245-0. PMID 8942565
- [Background] Caudle RJ, Stern PJ. Severe open fractures of the tibia. J Bone Joint Surg Am. 1987 Jul;69(6):801-7. PMID 3597491
- [Background] Madhuchandra P, Rafi M, Devadoss S, Devadoss A. Predictability of salvage and outcome of Gustilo and Anderson type-IIIA and type-IIIB open tibial fractures using Ganga Hospital Scoring system. Injury. 2015 Feb;46(2):282-7. doi: 10.1016/j.injury.2014.11.003. Epub 2014 Nov 15. PMID 25482348